CLINICAL TRIAL: NCT01145950
Title: A Randomized, Double-blind, Single-dosing, 2-way Cross-over Study to Compare the Safety and Pharmacokinetic Characteristics of LBEC0101 25 mg With Those of Enbrel® Injection 25 mg After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: Study to Compare the Safety and Pharmacokinetic Characteristics of LBEC0101 25 mg With Those of Enbrel®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Kim, Sung Il / Assistant Manager, Clinical Trial Team
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: LG-ECCL001
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Etanercept; Enbrel; healthy volunteers
MeSH Terms: interventions — LBEC0101; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: LBEC0101
- Group 2 (Experimental)
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: LBEC0101 — Etanercept 25mg, single dose
  Arms: Group 1
Drug: Enbrel — Etanercept 25mg, single dose
  Arms: Group 2

SUMMARY:
To compare the pharmacokinetic characteristic of LBEC0101 25mg with the active comparator, Enbrel® 25 mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 20 to 45 years of age the moment of screening
* Body mass index is between 18.0 and 30.0 kg/m

Exclusion Criteria:

* The tuberculosis patient or latent tuberculosis patient
* Hypersensitivity response to the test and comparator drugs

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Etanercept levels in blood | 22 day

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea